CLINICAL TRIAL: NCT06895408
Title: Separate and Combined Extrapancreatic Effects of Glucose-dependent Insulinotropic Polypeptide (GIP) and Glucagon-Like Peptide 1 (GLP-1)
Brief Title: Separate and Combined Extrapancreatic Effects of GIP and GLP-1
Acronym: GA-19b
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Asger Lund, MD, Clinical Associate Professor, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 101292 (H-21035117)
Record Dates: First submitted 2025-03-17; First posted 2025-03-26 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Pancreatectomy; Hyperglycemia
MeSH Terms: conditions — Hyperglycemia | interventions — Infusions, Intravenous

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- GIP (Experimental): Intravenous infusion of glucose-dependent insulinotropic polypeptide
  Interventions: Other: Intravenous Infusion
- GLP-1 (Experimental): Intravenous infusion of glucagon-like peptide 1
  Interventions: Other: Intravenous Infusion
- GIP + GLP-1 (Experimental): Intravenous infusion of glucose-dependent insulinotropic polypeptide and glucagon-like peptide 1
  Interventions: Other: Intravenous Infusion
- Saline (Placebo Comparator): Intravenous infusion of saline
  Interventions: Other: Intravenous Infusion

INTERVENTIONS:
Other: Intravenous Infusion — Glucose-dependent Insulinotropic Polypeptide
  Arms: GIP
Other: Intravenous Infusion — Glucagon-Like Peptide 1
  Arms: GLP-1
Other: Intravenous Infusion — Glucose-dependent Insulinotropic Polypeptide and Glucagon-Like Peptide 1
  Arms: GIP + GLP-1
Other: Intravenous Infusion — Saline
  Arms: Saline

SUMMARY:
The two gut-derived hormones, glucose-dependent insulinotropic polypeptide (GIP) and glucagon-like peptide 1 (GLP-1) are secreted from intestinal cells in relation to a meal and increase insulin secretion from the pancreas. The hormones also exert effects outside the pancreas, but especially for GIP, these are poorly investigated. Because of this, only GLP-1 based drugs (GLP-1 receptor agonists) are on the market for the treatment of type 2 diabetes and obesity. Nonetheless, a new drug is in clinical development: a combined GIP-GLP-1-receptor agonist (tirzepatide), which has shown better results than GLP-1 alone. The mechanism behind these impressive effects are unknown and in this study, the investigators will look into the exptrapancreatic effects of GIP and GLP-1, separate and combined and thus elucidate the mechanisms of action of this new drug class.

ELIGIBILITY:
Inclusion Criteria:

* Total pancreatectomy
* Caucasians between 30-75 years of age
* Blood haemoglobin >7.0 mmol/l for males and >6.5 mmol/l for females

Exclusion Criteria:

* Pancreatectomy within the last 3 months
* Ongoing chemotherapy or chemotherapy within the last 3 months
* Treatment with GLP-1 receptor agonists within the last 3 months
* Renal impairment (estimated by estimated glomerular filtration rate (eGFR) <60 ml/min/1.73 m2) and/or albuminuria
* Calcium related disease, hypo-/hyperthyroidism
* Known significant liver disease, plasma alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥3 × normal value or INR (The international normalised ratio based on prothrombin time) outside the normal range
* Severe arteriosclerotic heart disease or heart failure (New York Heart Association (NYHA) group III or IV)
* Pregnancy and/or breastfeeding
* Use of more than 14 units of alcohol per week or abuse of narcotics
* Any condition that the investigator feels would interfere with trial participation

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2025-02-19 (Actual); Primary Completion 2025-07-14 (Actual); Study Completion 2025-07-14 (Actual)

PRIMARY OUTCOMES:
Plasma glucose | Up to two months
  Changes in plasma levels of glucose between interventions assessed through frequently blood sampling during the experimental days
Plasma glucagon | Up to two months
  Changes in plasma levels of glucagon (gut-derived) between interventions assessed through frequently blood sampling during the experimental days
Plasma Insulin/C-peptide | Up to two months
  Changes in plasma levels of insulin/C-peptide between interventions assessed through frequently blood sampling during the experimental days
Plasma triglycerides | Up to two months
  Changes in plasma triglycerides between interventions assessed through frequently blood sampling during the experimental days
Plasma CTX | Up to two months
  Changes in CTX between interventions assessed through frequently blood sampling during the experimental days
Plasma PINP | Up to two months
  Changes in plasma PINP between interventions assessed through frequently blood sampling during the experimental days

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Clinical Metabolic Research, Gentofte Hospital, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: Undecided